CLINICAL TRIAL: NCT03467386
Title: Pilot Study of Total Marrow/Lymphoid Irradiation (TMLI) Conditioning Prior to Allogeneic Hematopoietic Stem Cell Transplant (HCT) Followed by Post Transplant Cyclophosphamide-Based Graft Versus Host Disease Prophylaxis for Acute Myelogenous Leukemia in Complete Remission
Brief Title: Total Marrow and Lymphoid Irradiation Before Donor Transplant and Cyclophosphamide in Treating Patients With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17423; NCI-2018-00177 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17423 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2018-02-22; First posted 2018-03-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Stem Cell Transplantation; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (TMLI, cyclophosphamide) (Experimental): Patients undergo TMLI BID on days -4 to 0, then undergo bone marrow or peripheral blood stem cell transplant on day 0. Patients receive cyclophosphamide IV over 2 hours on days 3 and 4, tacrolimus given by CIV on days 5-90, and filgrastim beginning on day 5 until ANC is at least 1,500/mm^3 for 3 consecutive days.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tacrolimus; Radiation: Total Marrow Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo alloHCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim — Administer according to City of Hope standard operating procedures
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Tacrolimus — Given CIV
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total Marrow Irradiation — Undergo TMLI

SUMMARY:
This pilot phase I trial studies the side effects of total bone marrow and lymphoid irradiation and how well it works with cyclophosphamide in treating patients with acute myeloid leukemia. Total marrow and lymphoid irradiation targets cancer in bone marrow and blood, instead of applying radiation to the whole body. Giving total bone marrow and lymphoid irradiation before a donor transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving total bone marrow and lymphoid irradiation before donor transplant and cyclophosphamide after transplant may work better at treating acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety/feasibility of combining a total marrow and lymphoid irradiation (TMLI) transplant conditioning regimen with a post-transplant high dose cyclophosphamide (PTCy)-based graft versus host disease (GvHD) prophylaxis strategy, through the assessment of: adverse events: type, frequency, severity, attribution, time course, duration and complications: including acute GvHD, infection and delayed neutrophil/platelet engraftment.

SECONDARY OBJECTIVES:

I. To estimate the cumulative incidence (CI) of acute GvHD at 100 days post allogeneic hematopoietic cell transplantation (alloHCT).

II. To estimate the CI of chronic GvHD at 6 months, 1- and 2-years post alloHCT.

III. To estimate GVHD-free relapse-free survival (GRFS) at 1- and 2-years post alloHCT.

IV. To describe the kinetics of immune reconstitution and T cell repertoire in the first year post alloHCT.

V. To estimate overall survival (OS), relapse-free survival (RFS) and CI of relapse, and non-relapse mortality (NRM) at 100 days, 1- and 2-years post alloHCT.

VI. To characterize quality of life using 36-Item Short Form Health Survey (SF-36), Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT), and M. D. Anderson Symptom Inventory (MDASI) or Pediatric Quality of Life Inventory (PedsQL) at 100 days, 6 months, 1- and 2-years post alloHCT.

VII. To assess bone marrow cellularity from bone marrow samples. VIII. To assess the clonogenic potential of cells from bone marrow samples. IX. To assess stromal damage from bone marrow samples. X. To evaluate cytokines and oxidative stress markers.

OUTLINE: This is a dose-escalation study of TMLI.

Patients undergo TMLI twice daily (BID) on days -4 to 0, then undergo bone marrow or peripheral blood stem cell transplant on day 0. Patients receive cyclophosphamide intravenously (IV) over 2 hours on days 3 and 4, tacrolimus given by continuous intravenous infusion (CIV) on days 5-90, and filgrastim beginning on day 5 until absolute neutrophil count (ANC) is at least 1,500/mm^3 for 3 consecutive days.

After completion of study treatment, patients are followed for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* This study is open to patients with acute myeloid leukemia (AML) evaluated within 30 days of the start of conditioning regimen and in first or second complete remission (CR)
* Karnofsky performance status (KPS) >= 70%
* The effects of radiation on the developing fetus are known to be teratogenic; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Patients with acute myelogenous leukemia (AML) who are in first or second complete remission
* All candidates for this study must have a human leukocyte antigen (HLA) (A, B, C, DR) identical sibling who is willing to donate primed blood stem cells (preferred) or bone marrow, or have a 10/10 allele matched unrelated donor; all ABO blood group combinations of the donor/recipient are acceptable since even major ABO compatibilities can be dealt with by various techniques; (red cell exchange or plasma exchange)
* A cardiac evaluation with an electrocardiogram showing no ischemic changes or abnormal rhythm and an ejection fraction of >= 50% established by multi-gated acquisition scan (MUGA) or echocardiogram
* Patients must have a serum creatinine of less than or equal to 1.3 mg/dL or creatinine clearance > 70 ml/min as calculated by the Cockcroft-Gault formula
* A bilirubin of less than or equal to 1.5 mg/dL, excluding patients with Gilbert's disease
* Patients should also have a serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) less than 5 times the upper limit of normal
* Pulmonary function tests including diffusing capacity of the lung for carbon monoxide (DLCO) will be performed; forced expiratory volume in 1 second (FEV 1) and DLCO should be greater than 50% of predicted normal value
* All subjects must have the ability to understand and the willingness to sign a written informed consent; signed informed consent form approved by the Institutional Review Board (IRB) is required; the patient, family member, and transplant staff physician (physician, nurse, and social worker) meet at least once prior to starting the transplant procedure; during this meeting, all pertinent information with respect to risks and benefits to the donor and recipient will be presented; alternative treatment modalities will be discussed
* The time from the end of last induction, re-induction, or consolidation regimen should be greater than or equal to 14 days
* Prior therapy with etoposide and cyclophosphamide is allowed
* DONOR: donor evaluation and eligibility will be assessed as per current City of Hope standard operating procedure (SOP)

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active or poorly controlled infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy; maintenance therapy with Food and Drug Administration (FDA)-approved targeted therapies (e.g. tyrosine kinase inhibitors for Philadelphia chromosome [Ph] positive [+] acute lymphoblastic leukemia [ALL], and FLT inhibitors for FLT3+ patients) will be allowed after day 60 disease assessment
* Prior radiation therapy that would exclude the use of TMLI
* Relapsed patients who have undergone autologous or allogeneic hematopoietic stem cell transplantation previously
* Patients with psychological or medical condition that patient's physician deems unacceptable to proceed to allogeneic hematopoietic stem cell transplantation
* Electrocardiogram (EKG) showing ischemic changes or abnormal rhythm and/or an echocardiogram or MUGA scan showing abnormal wall motion or ejection fraction < 50%
* Patients who have been treated with chemotherapy or radiation for the purpose of induction, re-induction or consolidation, within two weeks of planned study enrollment
* Patients with other active malignancies are ineligible for this study, other than localized malignancies
* Patients that are pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, including but not limited to, infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
1a. Incidence of adverse events | Up to 24 months
  Assessed using Bearman Scale Regimen-Related Toxicity scale. Scale range: Grade 0-4 (increasing grade reflects increasing severity), where Grade 0-none/did not experience and Grade 4=death.
1b. Incidence of adverse events | Up to 24 months
  Assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale. Scale range: Grade 1-5 (increasing grade reflects increasing severity), where Grade 1 reflects a more milder form of the adverse event and Grade 5=death.

SECONDARY OUTCOMES:
Time to neutrophil and platelet recovery/engraftment | From day 0 to recovery or declaration of engraftment failure, assessed up to 24 months
Acute graft versus host disease (GvHD) | Day 0 to 100 (120) days post-transplant
  Graded according to the Consensus Grading. The first day of acute GvHD onset at a certain grade will be used to calculate cumulative incidence curves for that GvHD grade; relapse/death prior to onset will be considered competing events. Will be calculated using the competing risk method as described by Gooley et al. (1999).
Chronic GVHD | From day (80) 100 to the onset of chronic GvHD, death or last contact, whichever comes first, assessed up to 24 months
  The first day of chronic GvHD onset will be used to calculate cumulative incidence curves, with relapse/death prior to onset considered competing events. Will be calculated using the competing risk method as described by Gooley et al. (1999).
GvHD-free/relapse-free survival (GRFS) | From start of treatment (hematopoietic stem cell transplant [HCT]) to grade 3-4 acute GvHD, chronic GvHD requiring systemic treatment, relapse, or death (from any cause), whichever occurs first, assessed p to 24 months
  Will be calculated using the Kaplan-Meier method.
Levels of immune cells | Up to 24 months
  Will be measured by flow cytometry for cell subsets: a. T-cells.
Levels of immune cells | Up to 24 months
  Will be measured by flow cytometry for cell subsets: b. B-cells.
Levels of immune cells | Up to 24 months
  Will be measured by flow cytometry for cell subsets: c. natural killer (NK) cells.
Levels of immune cells | Up to 24 months
  Will be measured by flow cytometry for cell subsets: d. regulatory T cells (T-regs).
Overall survival | From start of treatment until death, or last follow-up, whichever comes first, assessed up to 24 months
  Will be calculated using the Kaplan-Meier method.
Relapse-free survival | From the start of treatment to the date of death, disease relapse, or last follow-up whichever occurs first, assessed up to 24 months
  Will be calculated using the Kaplan-Meier method.
Relapse | From start of therapy, assessed up to 24 months
  Will be calculated using the competing risk method as described by Gooley et al. (1999).
Non-relapse mortality (NRM) | From start of treatment until non-disease related death, or last follow-up, whichever comes first, assessed up to 24 months
  The cumulative incidence of NRM will be calculated reflecting relapse as a competing risk. Will be calculated using the Kaplan-Meier method and the competing risk method as described by Gooley et al. (1999).
Quality of life -Questionnaire | Up to 24 months
  Assessed using a. 36-Item Short Form Health Survey (SF-36). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  * a1. vitality
  * a2. physical functioning
  * a3. bodily pain
  * a4. general health perceptions
  * a5. physical role functioning
  * a6. emotional role functioning
  * a7. social role functioning
  * a8. mental health
Quality of life-Function Assessment | Up to 24 months
  Assessed using b. Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT). (FACT-BMT) is a 47-item, valid and reliable measure of five dimensions of quality of life in bone marrow transplant patients. The dimensions collected and assessed are:
  * b1.physical well being
  * b2. Social and family well being
  * b3. Emotional well being
  * b4. Functional well being
  * b5. Additional concerns.
Quality of life -Symptom Inventory | Up to 24 months
  Assessed using c. M. D. Anderson Symptom Inventory (MDASI). MDASI is a multi-symptom patient-reported outcome (PRO) measure for clinical and research use. Use the MDASI to assess the severity of symptoms experienced by patients with cancer and the interference with daily living caused by these symptoms. The following parameters will be reported:
  * c1a. Pain
  * c1b. Fatigue
  * c1c. Nausea
  * c1d. Disturbed sleep
  * c1e. Distress/feeling upset
  * c1f. Shortness of breath
  * c1g. Difficulty remembering
  * c1h. Lack of appetite
  * c1i. Drowsiness
  * c1j. Dry mouth
  * c1k. Sadness
  * c1l. Vomiting
  * c1m. Numbness/tingling
  * c1n. Walking
  * c1o. Activity
  * c1p. Working (including housework)
  * c1q. Relations with other people
  * c1r. Enjoyment of life
  * c1s. Mood A total of eight quality of life parameters will be reported on each pediatric transplant patient.
  * c2a.Pain and Hurt
  * c2b. Fatigue and Sleep
  * c2c. Nausea
  * c2d. Worry
  * c2e. Nutrition
  * c2f. Thinking
  * c2g. Communication
Bone marrow residual damage assessment | Up to 24 months
Cytokines | Up to 24 months
Oxidative stress Markers | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S Stein, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States